CLINICAL TRIAL: NCT03068858
Title: Real-time Feedback of SYNTAX Score Category During Coronary Angiographies to Improve Appropriateness of Coronary Revascularization for Patients With Stable Coronary Artery Diseases: a Before-and-after Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160826
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Syntax Score; Appropriateness; Coronary Revascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SYNTAX score category feedback group (Experimental): A real-time SYNTAX score category feedback from angiographic core lab will be given to the cardiologists rightafter the angiographies.
  Interventions: Diagnostic Test: real-time feedback of SYNTAX score category
- Controlled group (No Intervention): Cardiologists' subjective SYNTAX score category judgement will be recorded during the angiography.

INTERVENTIONS:
Diagnostic Test: real-time feedback of SYNTAX score category
  Arms: SYNTAX score category feedback group

SUMMARY:
The SYNTAX score (SS) has been recommended by clinical guideline and appropriate use criteria for coronary revascularization (CR) to provide guidance on optimal treatment strategies for patients with stable coronary artery diseases (CAD). However, discrepancy in SS between angiographic core lab (ACL) and cardiologists has been found. Whether the misestimate will lead to inappropriate CR and whether a SS intervention will improve CR appropriateness in patients with stable CAD remain unknown.

Thus, our study aims at evaluating whether a real-time feedback from ACL rightafter the angiographies will improve CR appropriateness. A before-and-after controlled trial was designed. In the first period of time, stable CAD patients undergoing elective coronary angiographies with at least one coronary lesion stenosis ≥ 50% from one Chinese cardiac center will be continuously recruited as the control group. In the second period, eligible patients will be recruited continuously and a real-time SS category feedback from ACL rightafter the angiography will be given to the cardiologists. Appropriateness of treatment strategies in two groups will be analyzed to determine whether a real-time SS feedback can improve the treatment appropriateness. The appropriateness of treatment strategies will be adjudicated by Chinese version appropriate use criteria for CR.

ELIGIBILITY:
Inclusion Criteria:

1. Undergo elective coronary angiography with at least one coronary lesion stenosis ≥ 50%;
2. Patients with stable coronary artery diseases (stable angina, no or non-ischemic symptom);
3. Written informed consent.

Exclusion Criteria:

1. Have prior CABG;
2. Have stage PCI;
3. Have no assigned scenario in Chinese appropriate use criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3245 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Inappropriate rate of coronary revascularization | 1 month after study completion
  Inappropriate rate will be adjudicated by Chinese appropriate use criteria for coronary revascularization.

SECONDARY OUTCOMES:
The proportion of inappropriate PCI | 1 month after study completion
  Inappropriate rate of percutaneous coronary intervention (PCI) will be adjudicated by Chinese appropriate use criteria for coronary revascularization.
The proportion of inappropriate CABG | 1 month after study completion
  Inappropriate rate of coronary artery bypass graft (CABG) will be adjudicated by Chinese appropriate use criteria for coronary revascularization.
The proportion of utilizing PCI procedures | 1 month after study completion
  The proportion of patients who undergo percutaneous coronary intervention (PCI) among total patients
The proportion of utilizing CABG procedures | 1 month after study completion
  The proportion of patients who undergo coronary artery bypass graft (CABG) among total patients

CONTACTS AND LOCATIONS:
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin S, Zhang H, Chen SP, Rao CF, Wu F, Zhou FJ, Wang Y, Yan HB, Dou KF, Wu YJ, Tang YD, Xie LH, Guan CD, Xu B, Zheng Z. Mis-estimation of coronary lesions and rectification by SYNTAX score feedback for coronary revascularization appropriateness. Chin Med J (Engl). 2020 Jun 5;133(11):1276-1284. doi: 10.1097/CM9.0000000000000827. PMID 32452896